CLINICAL TRIAL: NCT06037135
Title: The Effects of Perioperative Dexmedetomidine Infusion on Hemodynamic Stability During Laparoscopic Adrenalectomy for Pheochromocytoma: a Randomized Study
Brief Title: Dexmedetomidine Infusion During Laparoscopic Adrenalectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2012-0577
Record Dates: First submitted 2023-08-08; First posted 2023-09-14 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Pheochromocytoma
MeSH Terms: conditions — Pheochromocytoma | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine group (Experimental): In the dexmedetomidine group, dexmedetomidine is administered at a rate of 0.5 μg/kg/h immediately after anesthesia induction and continued until the completion of the surgery.
  Interventions: Drug: dexmedetomidine
- Control group (Active Comparator): In the control group, a 0.9% normal saline infusion is initiated at the same rate immediately after anesthesia induction and continued until the end of the operation.
  Interventions: Drug: 0.9% normal saline

INTERVENTIONS:
Drug: dexmedetomidine — In the dexmedetomidine group, dexmedetomidine is administered at a rate of 0.5 μg/kg/h immediately after anesthesia induction and continued until the completion of the surgery. The research nurse, who did not participate in the study other than the management and preparation of the study medication, prepared 50mL of 0.9% normal saline for the control group and a mixture of dexmedetomidine 2 mL and 0.9% normal saline 48 mL (at a concentration of 4 μg/mL) for the dexmedetomidine group.
  Arms: dexmedetomidine group
Drug: 0.9% normal saline — In the control group, a 0.9% normal saline infusion is initiated at the same rate immediately after anesthesia induction and continued until the end of the operation.
  Arms: Control group

SUMMARY:
The investigators planned this study to investigate the effects of dexmedetomidine administration on intraoperative hemodynamic stability in patients with pheochromocytoma.

ELIGIBILITY:
Inclusion Criteria:

1. ages of 20 and 70
2. American Society of Anesthesiologists(ASA) physical status classification I to III,
3. planned laparoscopic adrenalectomy for pheochromocytoma.

Exclusion Criteria:

1. emergency operation,
2. re-operation,
3. combined surgery with other departments,
4. body mass index (BMI) >32 kg/m2,
5. history of arrhythmias (especially AV nodal block) and ventricular conduction abnormalities,
6. uncontrolled hypertension (diastolic blood pressure >110mmHg)
7. bradycardia (heart rate < 40 beats per minute),
8. history of heart failure, hepatic and/or renal failure,
9. history of cerebrovascular disease (cerebral hemorrhage, cerebral ischemia),
10. history of beta-blocker therapy, 10) history of uncontrolled psychiatric disease.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12-03 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Intraoperative hemodynamic stability ( maximum blood pressure during surgery (systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MBP)) | during operation
Intraoperative hemodynamic stability (duration of SBP increase by 30% or more from baseline (in minutes) | during operation
Intraoperative hemodynamic stability (duration of SBP exceeding 200 mmHg) | during operation
Intraoperative hemodynamic stability (maximum HR during surgery) | during operation
Intraoperative hemodynamic stability (duration of HR exceeding 110 beats per minute during surgery) | during operation
Intraoperative hemodynamic stability (comparison of the quantity of vasoactive drugs (nitroprusside, esmolol, norepinephrine) used during surgery) | during operation

SECONDARY OUTCOMES:
levels of catecholamines | immediately after anesthesia induction
  the actual secretion levels of catecholamines, specifically epinephrine and norepinephrine, were measured at different time points
levels of catecholamines | immediately after removal of the pheochromocytoma
  the actual secretion levels of catecholamines, specifically epinephrine and norepinephrine, were measured at different time points
levels of catecholamines | immediately after the completion of surgery
  the actual secretion levels of catecholamines, specifically epinephrine and norepinephrine, were measured at different time points

CONTACTS AND LOCATIONS:
Overall Officials: Young Jun Oh, M.D., Ph.D., Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine
Locations (1):
- Severance hospital, Seoul, South Korea